CLINICAL TRIAL: NCT03256240
Title: Prospective Randomized Study of the Kono-S Anastomosis Versus the Side-to-side Functional End Anastomosis in the Prevention of Post-operative Recurrence of Crohn's Disease
Brief Title: Study of the Kono-S Anastomosis Versus the Side-to-side Functional End Anastomosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1303013645
Record Dates: First submitted 2014-08-05; First posted 2017-08-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Crohn's Disease
Keywords: Crohn's recurrence
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to undergo either the Kono-S anastomosis or the side-to-side functional end anastomosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- side-to-side functional end anastomosis (Active Comparator): side-to-side functional end anastomosis creation
  Interventions: Other: side-to-side functional end anastomosis
- Kono-S (Active Comparator): antimesenteric functional side-to-side handsewn anastomosis, known as the Kono-S anastomosis
  Interventions: Other: Kono-S analstomosis

INTERVENTIONS:
Other: side-to-side functional end anastomosis — type of anastomosis
  Arms: side-to-side functional end anastomosis
Other: Kono-S analstomosis — antimesenteric anastomosis
  Arms: Kono-S

SUMMARY:
This study proposes a randomized prospective study comparing the Kono-S anastomosis to the standard side-to-side anastomosis.This will be a multi-center randomized prospective trial. Patients with Crohn's ileitis or Crohn's ileocolitis requiring resection will be randomized to undergo either the Kono-S anastomosis or the side-to-side functional end anastomosis.

DETAILED DESCRIPTION:
Study Aim:

* The primary aim of this study is to compare the postoperative recurrence of CD using the Rutgeerts score at 3-6 months between the novel Kono-S anastomosis (Group1) and side-to-side functional end anastomosis (Group2) and surgical recurrence rate at 60 and 120 months between the groups.
* The secondary aim is to evaluate the postoperative recurrence of CD using the Rutgeerts score at 12-18, 60 and 120 months between the groups; time to surgical recurrence between Group1 and Group2 measured in months from the index surgery, yearly Crohn's disease surgical therapy impact using the Work Productivity and Activity Impairment (WPAI) questionnaire; yearly Health-Related Quality of Life using the Short Inflammatory Bowel Disease Questionnaire, to evaluate before surgery, and yearly after the surgery up 60 months the patient perception of illness measured by The Brief Illness Perception Questionnaire, (a 9-item questionnaire) score between the groups, to evaluate disease activity yearly using Harvey-Bradshaw Index and monitor medication therapy, readmission rates, and mortality rates through the 60 months follow-up, and utilize Focus Groups from national and international study sites to evaluate patient's perspectives on surgical treatment, patients' goals of surgical treatment, and surgical treatment's personal and social impacts, patient perspective on nutrition; and caregiver perspective on surgical treatment, to evaluate histologic predictors for endoscopic and clinical remission in Crohn's Disease after ileocecal resection using the histological scores from the surgical pathology margin evaluation, to evaluate the differences in the histological mucosal healing between Kono-S and Side- to Side anastomosis measured by the histological score between the groups using the modified Global Histology Activity Score (Modified) between the groups

Methods

Design: This will be a multi-center randomized prospective trial with 500 subjects. Patients with Crohn's ileitis or Crohn's ileocolitis requiring initial resection will be randomized to undergo either the Kono-S anastomosis or the side-to-side functional end anastomosis.

Patients will be randomized into two Groups:

Group 1: Kono-S anastomosis vs. Group 2: side-to-side functional end anastomosis.

The purpose of this study is to compare the postoperative recurrence of Crohn's disease between the Kono-S procedure and the side-to-side functional end anastomosis and to evaluate the surgical recurrence rate at 60 and 120 months between the groups.

In any intestine surgery, after the sick portion of the bowel is removed, the intestinal tract is restored by reconnecting the healthy ends together. The new connecting line is called anastomosis and could be created in a variety of ways by the surgeon. This study will compare two different intestinal connections called Kono-S anastomosis and the traditional side-to-side functional end anastomosis. Initial studies have demonstrated that the Kono-S anastomosis has prevented endoscopic evidence of the post-operative recurrence of Crohn's disease at greater rates than the traditional side-to-side functional end anastomosis.

Follow-up: Patients will be discharged on no prophylactic treatments, and they will be followed post-operatively at 3 to 6, 12 to 18, 60-, and 120 months with a colonoscopy to assess for endoscopic recurrence. The mucosa will be graded with the Rutgeerts score for postoperative recurrence. All colonoscopies are part of the standard treatment. All patients will have also standard 30 days, 3 to 6, 12 to 18, 24, 36-, 48-, 60-, 72-, 84-, 96-, 108-, and 120 months follow-ups by phone call, through medical records, or during the postoperative clinic visit.

Follow-up Care: Patients with a Rutgeerts score at 3-to-6 months of:

* 0, 1, or 2a will be followed prospectively with or without introducing medical treatment at the discretion of the gastroenterologist.
* above >2a will initiate medical therapy for Crohn's disease
* Should the patient's symptoms warrant, medical treatment can be initiated at any time at the discretion of the gastroenterologist. This is a standard of care
* Colonoscopic images (still color photos acceptable) will be shown to a gastroenterologist blinded to the goal of the study for determination of the Rutgeerts score in addition to the initial evaluation by the sites endoscopists.
* post-operative endoscopic recurrence of CD using the Rutgeerts score at 12-18-, 60-, and 120 months between the groups. An endoscopic Rutgeerts score of 2b or higher will be considered a recurrence.
* Time to surgical recurrence between Group1 and Group2 measured in months from the index surgery
* Work Productivity and Activity Impairment (WPAI) questionnaire (a 6-item questionnaire that measures the amount of absenteeism and presenteeism due to health problems) will be administered annually for up to 120 months.
* Health-Related Quality of Life using the Short Inflammatory Bowel Disease Questionnaire (SIBDQ) (a 10-item shortened version of the original IBDQ, measuring the quality of life in four domains: bowel symptoms, emotional health, systemic systems, and social function) will be administered annually for up to 120 months.
* The Brief Illness Perception Questionnaire, (a 9-item questionnaire) score measuring the patient perception of illness before surgery, at 24-, 36-, 48-, 60-, 72-, 84-, 96-, 108-, and 120-months post-procedure.
* Harvey Bradshaw Index as a marker of clinical disease activity will be used. This will be recorded before the procedure (baseline), at 3 to 6 and 12-18 months, 24-, 36-, 48-, 60-, 72-, 84-, 96-, 108-, and 120-months post-procedure.
* Other monitoring- monitor medication therapy, readmission rates, and mortality rates annually through the 60 months of follow-up between the groups
* Focus groups from national and international study sites to evaluate patients' perspectives on surgical treatment, patients' goals of surgical treatment, and surgical treatment's personal and social impacts, patient perspective on nutrition; and caregiver perspective on surgical treatment. This is a qualitative evaluation.
* surgical pathology margin evaluation will be used to assess for histologic predictors for endoscopic and clinical remission in Crohn's Disease after ileocecal resection
* The differences in the histological mucosal healing between Kono-S and Side- to Side anastomosis measured by the histological score between the groups using the modified Global Histology Activity Score (Modified) between the groups at 60 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Crohn's ileitis or ileocolitis requiring initial surgical resection.
2. Age of 18 years and older, male and female
3. All Phenotypes of Crohn's diisease will be included: nonpenetrating (B1), stricturing (B2), and penetrating (fistulating) (B3), according to the Vienna classification
4. The patients can be on any medications coming into surgery, including prior anti- tumor necrosis factor(TNF) therapy.

Exclusion Criteria:

1. Patients under 18 years of age
2. Patients with recurrent Crohn's
3. Pregnant patients
4. Patients with more than one non-contiguous site of active disease, thus requiring multiple resections or additional bowel sparing procedures at the time of surgery.
5. Patients with Crohn's disease extending to the cecum and ascending colon
6. Patients who will need preventive postoperative medical treatment
7. Patients that need change of surgical procedure as per the surgeon at the time of the intraoperative abdominal evaluation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-03-12 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative remission of Crohn's disease between 3 and 6 months after surgery | 3-6 months after surgery
  Endoscopic remission with a Rutgeert score between 3 and 6 months in order to determine if the Kono-S procedure is more likely to prevent post-operative recurrence of Crohn's disease compared with the side-to-side functional end anastomosis. Endoscopic remission is defined as a Rutgeerts score of 0, 1, or 2a at 3-to-6 months post-procedure colonoscopy.
Number of subjects with surgical recurrence at 60 months | 60 months after surgery
  Number of anastomoses in need of surgical revision for Crohn's disease recurrence after the initial index surgery.
Number of subjects with surgical recurrence at 120 months | 120 months after surgery
  Number of anastomoses in need of surgical revision for Crohn's disease recurrence after the initial index surgery.

SECONDARY OUTCOMES:
Post-operative remission of Crohn's disease between 12 and 18 months, at 60-, and 120 months after surgery | 12-18, 60, and 120 months after surgery
  Endoscopic remission with a Rutgeerts score at 12 to 18, 60-, and 120 months in order to determine if the Kono-S procedure is more likely to prevent post-operative recurrence of Crohn's disease compared with the side-to-side functional end anastomosis. An endoscopic Rutgeerts score of 2b or higher will be considered a recurrence.
Work Productivity and Activity Impairment (WPAI) due to Crohn's disease | up to 120 months
  Work Productivity and Activity Impairment (WPAI) is a validated 6-item questionnaire that measures the amount of absenteeism and presenteeism due to CD during and activity impairment the 7 days prior to administration. It consists of 6 questions with the following domains: 1) employment status; 2) hours missed due to CD; 3) hours missed due to other reasons; 4) hours actually worked; 5) the degree to which CD affected productivity while working from 0 (no effect) to 10 (maximum impairment); and 6) the degree to which CD affected regular activities from 0 (no effect) to 10 maximum impairment ). All six question' domains will be reported and compared between the groups. Between the groups and within patients, changes will be evaluated. The mean score annual variability in each domain will be evaluated.
Health-Related Quality of Life using the Short Inflammatory Bowel Disease Questionnaire for Crohn's disease(10 questions) | up to 120 months
  Validated questionnaire to evaluate the quality of life in IBD patients. The short Inflammatory Bowel Disease Questionnaire (SIBDQ) is a 10-item shortened version of the original IBDQ, which was 32 items. Measures quality of life as measured in four domains, bowel symptoms, emotional health, systemic systems, and social function. SIBDQ score ranges between 10 and 70 points. QUOL is considered to be slightly (60-70 points), moderately (45-60 points), or severely impaired (10-45 points). In our study, the cut-off for relevant impairment of QUOL < 60 points.
Clinical disease activity measured by Harvey Bradshaw Index | up to 120 months
  Harvey Bradshaw Index is a marker of clinical disease activity. The following score grading system will be used to determine the clinical disease activity:
  Remission < 5 Mild disease 5-7 Moderate disease 8-16 Severe disease >16
Time to surgical recurrence between Group1 and Group2 | up to 120 months
  Time to surgical recurrence between Group1 and Group2 measured in months from the index surgery
Focus Group | up to 120 months
  Patient Focus Groups from national and international study sites to evaluate patient's perspectives on surgical treatment, patients' goals of surgical treatment, and surgical treatment's personal and social impacts, patient perspective on nutrition, and caregiver perspective on surgical treatment.
Medication therapy type | up to 120 months
  Medication therapy for Crohn's disease after the index surgery. We will monitor the type of medications patients receive after surgery. The following five types of medications will be recorded: Biologics, Immunosuppressants, Corticosteroids, Anti-Inflammatory, and Antibiotics.
Readmission rates between Group1 and Group2 | up to 120 months
  Number of readmission due to Crohn's disease after the index surgery
Mortality rate | up to 120 months
  Number of patient expired after the index surgery
Surgical Pathology Margins | at surgery
  Histological evaluation of the surgical pathology margin evaluation for presence or absence of disease
Mucosal Healing | 60 months after surgery
  Mucosal Healing from colonoscopy biopsies using the modified Global Histology Activity Score (Modified) score between the groups. Global Histology Activity Score (GHAS) is a widely used tool that grades biopsies of the ileum and colonic segments. The score has 8 domains and includes the presence of architectural changes, degree of chronic, neutrophilic and eosinophilic inflammatory infiltration in lamina propria, presence of intraepithelial neutrophils, epithelial damage, mucosal defects, presence of granulomas, and the extent of inflammation (proportion of biopsy specimens affected). Each domain is scored independently, and the total score is the sum of all individual scores, ranging from 2 (being the lowest meaning no histological activity) to 16 (being the highest meaning high histological disease activity).
Mucosal Healing from colonoscopy biopsies | 60 months after surgery
  Mucosal Healing from colonoscopy biopsies using The Inflammatory Bowel Disease-Distribution, Chronicity, Activity [IBD-DCA] score between the groups. The score is validated and has 3 domains: 1) Distribution of the disease; 2) Chronicity of the disease; and 3) Activity of the disease. Each domain of the IBD-DCA is scored as one of 0 (normal), 1 (mild), or 2 (moderate to severe) based on the presence of established histological findings and the domains are separately reported.
  Distribution [D] 0=Normal
  1. < 50% of tissue affected per same biopsy site
  2. ≥ 50% of tissue affected per same biopsy site Chronic features [C] 0=Normal
  1=Crypt distortion and/or mild lymphoplasmacytosis 2=Marked lymphoplasmacytosis and/or marked basal plasmacytosis Activity features [A] 0=Normal
  1. Two or more neutrophils in lamina propria in one high-power field [HPF] and/or intraepithelial neutrophils [any number]
  2. Crypt abscesses, erosions, ulcers
The Brief Illness Perception Questionnaire | up to 120 months
  The Brief Illness Perception Questionnaire, (a 9-item questionnaire) score with the nine items rated on a scale from 0 (minimum) to 10 (maximum), with higher scores indicating a more threatening perception of the illness. The total score is calculated by summing the scores of all eight items, with a possible range of 0-80. Higher scores indicate worse illness perception.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Michelassi, MD, Principal Investigator — Weill Medical College of Cornell University; Koianka Trencheva, Dr.PH,BSN,MS, Study Director — Weill Medical College of Cornell University
Locations (15):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington
- University Clinics Gasthuisberg Herestraat, Leuven, Belgium
- Helsinki University Hospital, Helsinki, Helsinki, Finland
- Germany (3):
  - Universitätsklinik Würzburg, Würzburg, Wurzburg
  - Charité Campus Benjamin Franklin, Berlin
  - Theresien Hospital and St. Hedwigs Clinic gGmbH, Mannheim
- Italy (3):
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Florence
  - Humanitas University Hospital, Rozzano, Milan
  - Policlinico University Hospital, Naples
- Hospital Universitario Vall d'Hebron, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Kono T, Ashida T, Ebisawa Y, Chisato N, Okamoto K, Katsuno H, Maeda K, Fujiya M, Kohgo Y, Furukawa H. A new antimesenteric functional end-to-end handsewn anastomosis: surgical prevention of anastomotic recurrence in Crohn's disease. Dis Colon Rectum. 2011 May;54(5):586-92. doi: 10.1007/DCR.0b013e318208b90f. PMID 21471760
- [Background] Kono T, Fichera A. Kono-S anastomosis for Crohn's disease: narrative - a video vignette. Colorectal Dis. 2014 Oct;16(10):833. doi: 10.1111/codi.12722. No abstract available. PMID 25040294